CLINICAL TRIAL: NCT04694729
Title: Comparison of the Effectiveness of Different Telerehabilitation Approaches in Chronic Obstructive Pulmonary Patients
Brief Title: Telerehabilitation Approaches in Chronic Obstructive Pulmonary Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Nursima Bulut, Physiotherapist, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TeleCOPD
Record Dates: First submitted 2021-01-02; First posted 2021-01-05 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Telerehabilitation; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Videoconference-based
  Interventions: Other: videoconference-based
- control group (Experimental): Video-based
  Interventions: Other: video-based

INTERVENTIONS:
Other: videoconference-based — Exercises will be done 3 days a week for 6 weeks, with the help of a physiotherapist via video conference.
  Arms: study group
Other: video-based — The exercise video will be sent to the patients and they will do it 3 days a week for 6 weeks. The subjects will be asked to keep an exercise diary and the status of the diaries will be followed by calling once a week.
  Arms: control group

SUMMARY:
Pulmonary rehabilitation (PR) is a first-line management strategy in chronic obstructive pulmonary patients (COPD) as it reduces shortness of breath, increases exercise capacity, and improves health-related quality of life. However, 8-50% of patients referred to PR do not participate at all, while 10-32% of those who start do not complete the program. Barriers to participation and completion include difficulty in accessing the program, poor mobility, lack of transport, and travel costs. Telerehabilitation is defined as the provision of rehabilitation services through telecommunication technology, including telephone, internet and video conference communications between the patient and the healthcare provider. Different technologies (from phone to video conferencing) have been tested in patients with COPD to enhance daily activities, exercise training and walking prescription. All of them showed positive effects on exercise tolerance, dyspnea, physical activity and quality of life. However, there is no study about which telerehabilitation program is more effective on COPD patients. The aim of this study is to investigate which telerehabilitation approach is more effective in COPD.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with COPD (FEV1 / FVC <70% in the stable phase of the disease)
* Age > 18 years old
* Have the ability to use a smartphone

Exclusion Criteria:

* Musculoskeletal disorders that limit exercise
* Dizziness, significant sensory or motor impairments, dementia or terminal illnesses that prevent education
* Serious comorbidities such as unstable heart disease, irregular diabetes, known malignant disease, any other disease that makes the patient unsuitable for participation in the study.
* Incompatible patient
* Severe vision or hearing impairment
* Unwillingness or inability to follow the protocol
* Have had a COPD exacerbation in the previous 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
6 minute walk test(6MWT) | 6 week
Pulmonary function testing | 6 week

SECONDARY OUTCOMES:
30-Second Chair Stand Test | 6 week
Time Up and Go Test | 6 week
Copd Assessment Test | 6 week
St George's Respiratory Questionnaire | 6 week
Hospital Anxiety and Depression Scale | 6 week
Medical Research Council Scale | 6 week
Short Physical Performance Battery | 6 week
International Physical Activity Questionnaire-Short Form | 6 week
Static Lung Volumes | 6 week

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital, Istanbul, Turkey (Türkiye)